CLINICAL TRIAL: NCT04863443
Title: Nonlinear Elasticity Mapping of Breast Masses
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Azra Alizad, Principal Investigator, Mayo Clinic
Other Study IDs: 14-004964; R01CA195527 (NIH)
Record Dates: First submitted 2021-04-22; First posted 2021-04-28 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Breast Cancer
Keywords: Breast; Mass
MeSH Terms: conditions — Breast Neoplasms; Arachnodactyly | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: Ultrasound — ultrasound scanner to collect sonographic imaging data from the breast
  Other Names: Supersonics Aixplorer; Verasonics; Alpinion

SUMMARY:
This proposed technique, called "Nonlinear Elasticity Mapping (NEM)", is an innovative approach to estimate (i.e., linear and nonlinear) elasticity to provide complementary and relevant information for identification and characterization of breast masses.

The proposed technique includes imaging the (nonlinear) elasticity parameter in a quantitative manner and measuring two new and relevant parameters. These parameters, together with linear elasticity, are used to differentiate breast masses. The first parameter is the nonlinearity of the elasticity.

DETAILED DESCRIPTION:
Measuring the nonlinearity of elasticity is obtained by recording ultrasound scans of object under different values of externally applied compression, and processing the resulting data. The central element of the proposed method is the solution of an inverse problem by which the linear and nonlinear parameters are estimated and a map of tissue nonlinearity is produced, in which the malignant masses can be identified. In addition to estimating the elasticity, will also evaluate the heterogeneity of the (linear) elasticity parameter distribution within the mass as an indicator of malignancy. In a previously performed pilot study, tested the proposed method on a small group of patients.

The goal of this project is to take the next logical step, which is to test this method in a clinical study on a larger population of patients to obtain statistically meaningful results. Assuming that the proposed method continues to demonstrate high specificity, this technique can have a significant impact on breast cancer diagnosis and management.

ELIGIBILITY:
Inclusion Criteria:

* Without a history of mastectomy or implants, which are identified to have findings on their clinical breast ultrasound.

Exclusion Criteria:

* Previous mastectomy or implants
* Any condition that does not allow proper use of imaging devices.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Female and male patient volunteers, aged 18 years and older, without a history of mastectomy or implants, which are identified to have findings on their clinical breast ultrasound
Sampling Method: Probability Sample
Enrollment: 172 (Actual)
Dates: Start 2014-07-24 (Actual); Primary Completion 2025-08-30 (Actual); Study Completion 2025-08-30 (Actual)

PRIMARY OUTCOMES:
Determine the diagnostic performance of the proposed nonlinear elasticity mapping method by measuring the nonlinear elasticity parameter. | Up to 2 weeks post breast biopsy
  In order to quantify this diagnostic potential we evaluate the average value of the relative shear modulus and the nonlinear parameter within each mass and correlate the results to the pathology results of breast biopsy.
Diagnostic performance of elasticity heterogeneity with measuring the combined linear and nonlinear elasticity parameters | Up to 2 weeks post biopsy
  Complement elasticity with additional quantitative information about linear and nonlinear elasticity parameters, that is relevant to the disease mechanism.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Mayo Clinic, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: Undecided